CLINICAL TRIAL: NCT00330538
Title: Incidence of Osteoporosis in Children With Acute Lymphoblastic Leukemia Undergoing Therapy
Brief Title: Osteoporosis in Children With ALL
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Other Study IDs: 03 08-085
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Leukemia, Lymphocytic, Acute, L1
Keywords: Osteoporosis; Childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Osteoporosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Hypothesis:

Pediatric patients with acute lymphoblastic leukemia, treated with chronic glucocorticoids as a part of the leukemia treatment protocol, will have an increased incidence and severity of osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is a disease characterized by low bone mass and microarchitectural deterioration of bone tissue. Osteoporosis is a devastating disorder with significant physical, psychosocial and financial consequences. Intensive chemotherapy and radiotherapy have led to significant improvements in long term, disease-free survival of children with malignancies. Unfortunately, there are many deleterious side effects associated with this therapy. Little is known about the longitudinal changes in bone mass accumulation and bone metabolism in these patients.

The purpose of this study is to evaluate the timing and severity of changes in bone mineral metabolism for children treated for childhood leukemia. Data will be used to establish treatment protocols with the goal of preventing severe fractures and pain in the acute treatment stage and severe osteoporosis and related pathology in the chronic stage.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients with a new diagnosis of ALL between ages 4-18
* Patients who are expected to receive glucocorticoids as part of the leukemia treatment protocol
* Bone density measurements must be performed at the diagnosis visit or maximally within 48 hours after the first dose of glucocorticoids

Exclusion Criteria:

* Patients under 4 years of age are excluded due to lack of age appropriate standards for bone mineral density
* Glucocorticoid therapy of at least one month or longer within the six months prior to DX
* History of connective tissue or musculoskeletal disorders
* Biphosphonate therapy within the past 6 months
* Acute renal failure
* Serum creatinine equal to or higher than 4.5mg/dl
* Positive serum pregnancy test in adolescent females

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2004-03; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jadranka Popovic, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States